CLINICAL TRIAL: NCT00189995
Title: Intramuscular Clozapine in the Management of Aggression in Schizophrenic Patients
Brief Title: Clozapine IM and Aggression in Schizophrenic Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Responsible Party: Principal Investigator, Vladimir Lerner, Associated Professor, Beersheva Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMHC-4000
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2005-10

CONDITIONS: Schizophrenia
Keywords: schizophrenia; aggression; clozapine; efficacy; double-blind
MeSH Terms: conditions — Schizophrenia; Aggression | interventions — Clozapine; Haloperidol

INTERVENTIONS:
Drug: clozapine
Drug: haloperidol

SUMMARY:
Aggressive, persistent aggression and impulsive behavior are frequently observed in schizophrenic patients. According to some researchers "more than 50% of all psychiatric patients and 10% of schizophrenic patients show aggressive symptoms varying from threatening behavior and agitation to assault"(1). It is a common cause of psychiatric admission and is a therapeutic issue. The treatment of these symptoms is a clinical problem for both patients and staff. Violent behavior, a major detrimental factor in stigmatization of the mentally ill, also poses physical danger for the patients themselves. Current pharmacotherapy of pathologic aggression involves the use of multiple agents (typical and atypical antipsychotics, benzodiazepines, mood stabilizers, beta-blockers, antiandrogenic hormones, and selective serotonin reuptake inhibitors) on empiric basis, with varying degrees of response (2-6). Unfortunately, these approaches lead to numerous side effects. Poor or noncompliance with pharmacotherapy makes it difficult to choose the appropriate preparation. Currently, typical neuroleptics are still the first choice in treating acute aggressive symptoms, while risperidone and olanzapine could be alternatives (5-7). Typical depot neuroleptics should be considered in cases where medication compliance is a problem. Most clinical information on treating of aggression has been collected about atypical neuroleptics, particularly regarding clozapine.

Clozapine is indicated in psychotic state and/or in drug-resistant schizophrenic patients. According to the FDA - it is the drug of choice in suicidal and aggressive patients, due-to psychotic state. It was found helpful in nearly 30% of resistant schizophrenic patients. Concerning the parenteral administration of clozapine - very little data is available today.

This study aims to investigate efficacy and safety (psychopathology, and side effects) of parenteral clozapine in treatment of aggressive behavior in schizophrenic patients in a double-blind trial.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenic, schizoaffective, or schizophreniform according to DSM-IV
* treatment-resistant
* presenting pathologic violent-aggressive behavior on admission
* at risk for self damage
* age: 18-65
* patient is not participating in any other study at time of this study
* minimal score of 70 on PANSS
* prior resistance to at least 2 different classes of neuroleptics
* OAS scores of at least 4 points in physical aggression sections and at least 2 points in verbal aggression section

Exclusion Criteria:

* neutropenia or any other abnormal CBC result
* myeloproliferative disease
* chronic physical diseases such as liver, renal or cardiac diseases
* history of alcohol or drug abuse
* history of drug induced granulocytopenia/agranulocytosis
* alcoholic/drug psychosis or intoxication
* carbamazepine or other bone marrow suppressor treatment
* uncontrolled epilepsy
* paralytic ileus
* hypersensitivity to clozapine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale
Overt Aggression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Valdimir Lerner, MD, PhD, Principal Investigator — Ben-Gurion University of the Negev; Baruch Spivak, MD, Principal Investigator — Tel Aviv University; Chanoch Midownik, MD, Principal Investigator — Ben-Gurion University of the Negev
Locations (2):
- Israel (2):
  - Beersheva Mental Health Center, Beersheva
  - Nes Ziona Medical Center, Ness Ziona